CLINICAL TRIAL: NCT00254891
Title: International, Randomized, Open-Label, Phase 3 Trial of Paclitaxel/Carboplatin Plus PF-3512676 Versus Paclitaxel/Carboplatin Alone as First-Line Treatment of Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Trial of Paclitaxel/Carboplatin + PF-3512676 vs Paclitaxel/Carboplatin Alone in Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Termination Reason in Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8501001
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: advanced carcinoma, non-small cell lung, Phase III, Paclitaxel, Taxol, Carboplatin, Paraplatin, PF-3512676, immunotherapy, immune modulator
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ProMune; Paclitaxel; Carboplatin; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Standard of care chemotherapy plus experiment intervention (PF-3512676)
  Interventions: Drug: PF-3512676 + Paclitaxel + Carboplatin
- B (Active Comparator): Standard of care chemotherapy
  Interventions: Drug: Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: PF-3512676 + Paclitaxel + Carboplatin — * PF-3512676: 0.2 mg/kg subcutaneously Days 8 and 15 of each 21 day cycle x 6 cycles then weekly as maintenance until disease progression or unacceptable toxicity.
  * Paclitaxel: 200 mg/m2 intravenously Day 1 of each 21 day cycle x 6 cycles.
  * Carboplatin: AUC 6 intravenously Day 1 of each 21 days cycle x 6 cycles.
  Other Names: Taxol; Paraplatin
  Arms: A
Drug: Paclitaxel + Carboplatin — * Paclitaxel: 200 mg/m2 intravenously Day 1 of each 21 day cycle x 6 cycles.
  * Carboplatin: AUC 6 intravenously Day 1 of each 21 days cycle x 6 cycles.
  Other Names: Taxol; Paraplatin
  Arms: B

SUMMARY:
To assess the efficacy and safety of PF-3512676 administered in combination with paclitaxel/carboplatin chemotherapy as first-line treatment in patients with locally advanced or metastatic Non-Small-Cell Lung Cancer (NSCLC) and to compare it to the efficacy and safety of paclitaxel

DETAILED DESCRIPTION:
PF-3512676 dosing was stopped 20 June 2007 in response to DSMC recommendation to close the trial, citing lack of efficacy concerns as the primary reason with a safety issue (sepsis) also contributing to the decision. Subjects were allowed to complete standard of care treatment/survival follow-up. Data collection was completed on 17 July 2008.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Non-Small-Cell Lung Cancer (NSCLC) stage IIIB with pleural effusion or stage IV
* No prior systemic treatment for Non-Small-Cell Lung Cancer (NSCLC)with chemotherapy, immunotherapy, biologic response modifiers or other investigational drugs
* Eastern Cooperative Oncology Performance Status (ECOG PS) 0 or 1

Exclusion Criteria:

* Small cell or carcinoid lung cancer
* Known Central Nervous System (CNS) metastasis
* Pre-existing auto-immune or antibody mediated diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2005-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 656 Events

SECONDARY OUTCOMES:
Overall Objective Response | End of Treatment
Time to Tumor Progression | Time of progressive disease
Progression Free Survival | Time of primary endpoint
Duration of Response | Time of progressive disease
Patient Reported Outcomes | End of Treatment
Overall Safety Profile | 28 days post PF-3512676 dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (165):
- United States (72):
  - Pfizer Investigational Site, Little Rock, Alaska
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Fayetteville, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Tucker, Georgia
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Jefferson, Indiana
  - Pfizer Investigational Site, New Albany, Indiana
  - Pfizer Investigational Site, Cedar Rapids, Iowa
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shelbyville, Kentucky
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Gretna, Louisiana
  - Pfizer Investigational Site, Lafayette, Louisiana
  - Pfizer Investigational Site, Marrero, Louisiana
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Biddeford, Maine
  - Pfizer Investigational Site, Brunswick, Maine
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Allegan, Michigan
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Saint Joseph, Michigan
  - Pfizer Investigational Site, Columbus, Mississippi
  - Pfizer Investigational Site, Corinth, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Papillion, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Ruidoso, New Mexico
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Great Neck, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Brevard, North Carolina
  - Pfizer Investigational Site, Lexington, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Dover, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Langhorne, Pennsylvania
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Arlington, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Richardson, Texas
  - Pfizer Investigational Site, Trophy Club, Texas
  - Pfizer Investigational Site, Bountiful, Utah
  - Pfizer Investigational Site, Layton, Utah
  - Pfizer Investigational Site, Murray, Utah
  - Pfizer Investigational Site, Provo, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, WVC, Utah
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Kennewick, Washington
  - Pfizer Investigational Site, Richland, Washington
  - Pfizer Investigational Site, Madison, Wisconsin
- Australia (12):
  - Pfizer Investigational Site, Albury, New South Wales
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Randwick, New South Wales
  - Pfizer Investigational Site, Pimlico, Queensland
  - Pfizer Investigational Site, Townsville, Queensland
  - Pfizer Investigational Site, Woolloongabba, Queensland
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, Toorak Gardens, South Australia
  - Pfizer Investigational Site, East Melbourne, Victoria
  - Pfizer Investigational Site, East Ringwood, Victoria
  - Pfizer Investigational Site, Wodonga, Victoria
  - Pfizer Investigational Site, Nedlands, Western Australia
- Belgium (2):
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Liège
- Canada (4):
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Rimouski, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- China (3):
  - Pfizer Investigational Site, Dalian, Xigang District, Liaoning
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai
- Pfizer Investigational Site, Nicosia, Cyprus
- Czechia (3):
  - Pfizer Investigational Site, Nová Ves pod Pleší
  - Pfizer Investigational Site, Ostrava-Poruba
  - Pfizer Investigational Site, Ústí nad Labem
- France (10):
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Herblain
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
- Germany (7):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bielefeld
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, München
- Greece (5):
  - Pfizer Investigational Site, Athens, Attica
  - Pfizer Investigational Site, Heraklion, Crete
  - Pfizer Investigational Site, Thessaloniki, Macedonia
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Rio, Patras
- Pfizer Investigational Site, Pokfulam, Hong Kong
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Debrecen
- India (5):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Chandigarh, Punjab
  - Pfizer Investigational Site, Jaipur, Rajasthan
- Pfizer Investigational Site, Ẕerifin, Israel
- Italy (4):
  - Pfizer Investigational Site, Lido Di Camaiore (LU)
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Pavia
- Mexico (2):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Puebla City, Puebla
- Netherlands (4):
  - Pfizer Investigational Site, Tiel, Gelderland
  - Pfizer Investigational Site, Groningen, Provincie Groningen
  - Pfizer Investigational Site, Amstelveen
  - Pfizer Investigational Site, The Hague
- Poland (2):
  - Pfizer Investigational Site, Otwock
  - Pfizer Investigational Site, Wodzislaw Sl.
- Portugal (3):
  - Pfizer Investigational Site, Faro
  - Pfizer Investigational Site, Porto
  - Pfizer Investigational Site, Vila Nova de Gaia
- South Africa (3):
  - Pfizer Investigational Site, Parktown, Gauteng
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Johannesburg
- Pfizer Investigational Site, Seoul, South Korea
- Spain (7):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Alcorcón, Madrid
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Pamplona, Navarre
  - Pfizer Investigational Site, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Madrid
- Sweden (2):
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uppsala
- Pfizer Investigational Site, Lausanne, Switzerland
- Pfizer Investigational Site, Taipei, Taiwan
- United Kingdom (7):
  - Pfizer Investigational Site, Truro, Cornwall
  - Pfizer Investigational Site, Exeter, Devon
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Portsmouth
  - Pfizer Investigational Site, Sheffield
  - Pfizer Investigational Site, Surrey GU2 5XX
  - Pfizer Investigational Site, Swansea

REFERENCES:
- [Derived] Roeland EJ, Fintelmann FJ, Yang R, Tarasenko L, Bonomi PD. Evaluation of Weight Gain and Overall Survival of Men Versus Women With Advanced Non-Small Cell Lung Cancer. J Cachexia Sarcopenia Muscle. 2025 Dec;16(6):e70131. doi: 10.1002/jcsm.70131. PMID 41332393
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8501001&StudyName=Trial%20of%20paclitaxel/carboplatin%20+%20PF-3512676%20vs%20paclitaxel/carboplatin%20alone%20in%20patients%20with%20advanced%20Non-Small%20Cell%20Lung%20Cancer%20